CLINICAL TRIAL: NCT05513131
Title: Clinical Study Protocol of Venetoclax Combined With Azacitidine and Harringtonine in the Treatment of Secondary Acute Myeloid Leukemia
Brief Title: Clinical Study Protocol of Venetoclax Combined With Azacitidine and Harringtonine in the Treatment of sAML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-376
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Secondary Acute Myeloid Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax combined with Azacitidine and Harringtonine (Experimental): Venetoclax 100mg d1，200mg d2，400mg d3~d14； Azacitidine 75mg/m2/d，d1~d7； Homoharringtonine 2mg/d d1~d7
  Interventions: Drug: Venetoclax；Azacitidine；Homoharringtonine

INTERVENTIONS:
Drug: Venetoclax；Azacitidine；Homoharringtonine — A cycle every 28 days Treatment with Venetoclax 100mg d1，200mg d2，400mg d3~d14； Azacitidine 75mg/m2/d，d1~d7 Homoharringtonine 2mg/d d1~d7

SUMMARY:
This research is being done to assess the therapeutic efficacy and safety of a promising regimen (Venetoclax combined with Azacitidine and Harringtonine) in patients with secondary AML

This study involves the following:

Venetoclax combined with Azacitidine and Harringtonine

DETAILED DESCRIPTION:
This is an open-label,single center, clinical trial to evaluate the efficacy and safety of Venetoclax in combination with Azacitidine and Harringtonine in patients with sAML

The FDA has approved the combination therapy of Venetoclax and Decitabine/Azacitidine for elderly (> 60-year-old) patients with newly diagnosed AML not eligible for intensive chemotherapy. Venetoclax is an inhibitor of BCL-2 (B-cell lymphoma 2, a protein that initiates tumor growth, disease progression, and drug resistance), which can lead to cancer cell death.

Homoharringtonine (HHT), a plant alkaloid with antitumor properties originally identified nearly 40 years ago, has a unique mechanism of action by preventing the initial elongation step of protein synthesis. HHT has been used widely in China for the treatment of chronic myeloid leukemia (CML), acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS)

Participants will receive 1-2 cycles of intensive treatment and followed with consolidated therapy with the same regimen of 4-6 cycles.If CR is not achieved by induction therapy, re-induction therapy can be continued, and those who have not achieved CR after re-induction therapy will withdraw from the study. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) if the patient meets the criteria for transplantation during treatment and a suitable donor exists After completion of study treatment, participants are followed up every 3 months for up to 2 years.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with acute myeloid leukemia (AML) newly diagnosed by bone marrow morphology and immunophenotyping (in line with the WHO 2016 diagnostic criteria), and meet any of the following conditions:

  * Patients with treatment-related AML (tAML);
  * AML patients with a previous history of MDS or CMML;
  * AML patients with myelodysplasia-related cytogenetic abnormalities; 2) Age ≥ 18 years old, and age < 80 years old; 3) Eastern Cooperative Oncology Group (ECOG) performance status score ≤2; 4) Aspartate aminotransferase (ALT), alanine aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 3 × upper limit of normal (ULN), serum bilirubin ≤ 1.5 × ULN; serum creatinine ≤ 2.0 × ULN; Serum myocardial enzyme <2.0×ULN; 5) LVEF determined by echocardiography ≥50%; Obtain informed consent signed by the patient or legal representative.

Exclusion Criteria:

* 1) AML with central nervous system (CNS) infiltration; 2) Acute promyelocytic leukemia confirmed by bone marrow morphology or immunophenotyping; 3) Have received Venetoclax treatment in the past; 4) Those who are known to be allergic to any drugs or other ingredients in the program; 5) Currently suffering from active autoimmune disease or a history of autoimmune disease potentially involving the CNS; 6) Known human immunodeficiency virus (HIV) infection; 7) Known history of active hepatitis B or C (HBV, HCV) infection; 8) Pregnant women and women who are trying to conceive; 9) Suffering from severe and/or uncontrolled mental illness; 10) Any life-threatening disease, health condition, or organ system dysfunction that the investigator believes may compromise the safety of the subject, or create an undue risk to the research results; 11) Received major surgery within 4 weeks before randomization; Participate in other clinical investigators at the same time one month before enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with complete remission (CR) and complete remission with incomplete marrow recovery (CRi) | From randomization to the end of Cycle 1 (each cycle is 28 days)
  CR is defined as absolute neutrophil count > 10^9/ L, platelets > 100×10^9/L, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of < 10^9/L or platelets < 100×10^9/L.

SECONDARY OUTCOMES:
Partial Remission (PR) Rate Secondary Outcome Measures: Secondary Outcome Measures: Partial Remission (PR) Rate | From randomization to the end of Cycle 1 (each cycle is 28 days)
  PR is defined as bone marrow with 5%~25% blasts, at least 50% lower than the initial diagnosis.
Overall Response Rate (ORR) | From randomization to the end of Cycle 1 (each cycle is 28 days）
  Complete Remission/ Complete Remission with incomplete count recovery/ Partial Remission/ Morphologic Leukemia Free State
Rate of Minimal Residual Disease (MRD) negativity | From randomization to the end of Cycle 1 (each cycle is 28 days)
  Percentage of participants who converted to MRD < 10^-3 before initiation of consolidation therapy. MRD is measured by MFC and RT-qPCR.
Overall survival (OS) | From the time of randomization to time for up to 2 years
  It is measured from the date of randomization to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Disease-Free Survival (DFS） | From the time of randomization to time for up to 2 years
  It is defined as the time from the date of CR/CRi to the date of recurrence or death.
The proportion of allogeneic hematopoietic stem cell transplantation | From the time of randomization to time for up to 2 years
  Proportion of allogeneic hematopoietic stem cell transplantation after disease remission
Cumulative incidence of relapse (CIR) | From the time of CR/CRi to time for up to 2 years
  It is measured from the date of CR/CRi to the date of relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No